CLINICAL TRIAL: NCT03280134
Title: CK19 Combined With Contrast-enhanced Ultrasound for Predicting Non-sentinel Lymph Node Status in Early Breast Cancer: a Prospectively Validation Cohort Study of the Predictive Model
Brief Title: A Prospective Validation Cohort Study of a Prediction System on nSLN Metastasis in Early Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, YU Xingfei, Dr., Zhejiang Cancer Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZJCH-CK19B
Record Dates: First submitted 2017-09-09; First posted 2017-09-12 (Actual); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Lymph Node Metastases; Breast Cancer; Predictive Cancer Model
Keywords: non-sentinel lymph node; breast cancer; prediction; CK19; contrast-enhanced ultrasound
MeSH Terms: conditions — Lymphatic Metastasis; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study based on prospective cohort method and concerning on the two groups (whether ALND or not) by predictive model nSLN results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- predictive nSLN- (No Intervention): No further axillary lymph node dissection (ALND)
- predictive nSLN+ (Active Comparator): axillary lymph node dissection (ALND)
  Interventions: Procedure: axillary lymph node dissection (ALND)

INTERVENTIONS:
Procedure: axillary lymph node dissection (ALND) — If the patients had predictive nSLN+, need further axillary lymph node dissection.
  Arms: predictive nSLN+

SUMMARY:
In the previous study, the investigator established a predictive model for non-sentinel lymph node involvement in early breast cancer (cT1-2cN0, 1-2 SLNs involvement). To validation the clinical value of the model, the investigator design a prospectively research using the model guiding for further axillary lymph node dissection in SLN-positve early breast cancer.

DETAILED DESCRIPTION:
In the previous study, a predictive model for non-sentinel lymph node involvement in early breast cancer (cT1-2cN0, 1-2 SLNs involvement) was established. This model was designed for predicting the status of non-sentinel lymph node in cT1-2cN0 with 1-2 SLNs involvement breast cancer based on peripheral blood CK19 and contrast-enhanced ultrasound. The investigator previously tested this model comparing with MSKCC model in a same population and confirmed a result of satisfactory low false-negative rate and high AUC. This model had a potential practise value in clinic applying. For further validation, the research group design the CK19B trial to prospectively using this model in decision strategy of whether receiving ALND in 1-2SLNs+ patients. If the model predictive result is negative, the risk of nSLNs involvement is estimated very low and the patients should be avoid ALND, even radiotherapy no matter the surgery is mastectomy or conserving. If the model result is positive, then further ALND or radiotherapy should be accepted by patients to decrease the risk of local and regional recurrent. A prospectively and conditional grouping method is planned for this cohort study. The primary endpoint is disease-free survival (DFS) in two groups, the second primary endpoint is local recurrent rate (LRR) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

the test group should be in accordance with the pathological diagnosis of breast cancer, the clinical stage of breast cancer (stage cTis, cI, cII and cT3N1M0), the initial treatment to receive surgical treatment. Complete preoperative clinical diagnosis data, including the ipsilateral axillary lymph node CEUS data and peripheral blood sample; The negative-control group should comply with the pathological diagnosis, breast adenosis, fibrocystic lesions, breast cysts and other benign lesions, with complete preoperative clinical data, also including ipsilateral axillary lymph node CEUS data and peripheral blood sample

Exclusion Criteria:

1. metastatic breast cancer, inflammatory breast disease, surgery without lymph node staging
2. pregnancy or lactation
3. patients with hematopoietic system disease or cancer, autoimmune diseases
4. preservation of substandard peripheral blood samples.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
disease-free survival (DFS) | 3-year(mid-term) 5-year
  The time from enrollment to the first recurrent or metastasis event

SECONDARY OUTCOMES:
local recurrent rate | 3-year(mid-term) 5-year
  The time from enrollment to the first time of local recurrent event (lymph drainage area recurrence)
overal survival (OS) | 3-year(mid-term) 5-year
  The time from enrollment to death for any reason

CONTACTS AND LOCATIONS:
Overall Officials: XF YU, M.D., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Qiao E, Yu X, Zhou L, Wang C, Yang C, Yu Y, Chen D, Huang J, Yang H. A Prospective Validation Cohort Study of a Prediction Model on Non-sentinel Lymph Node Involvement in Early Breast Cancer. Ann Surg Oncol. 2020 May;27(5):1653-1658. doi: 10.1245/s10434-019-07980-x. Epub 2019 Oct 28. PMID 31659631